CLINICAL TRIAL: NCT04561154
Title: Identifying Functional and Psycho-social Complaints After Hospitalization for Severe SARS-CoV-2 Infection (COVID19)- REPERCOV
Brief Title: Identifying Functional and Psycho-social Complaints After Hospitalization for SARS-CoV-2 Infection( COVID 19)- REPERCOV
Acronym: REPERCOV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHM-2020/S10/04
Record Dates: First submitted 2020-09-09; First posted 2020-09-23 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: SARS-COV2; COVID19
Keywords: SARS-COV2; functionnal complaints; sequel
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient hospitalized between march 1 and june 30, 2020 (Experimental): patient hospitalized between march 1 and june 30, 2020
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — three months after hospitalization, a questionnaire will be sent to patients. If necessary, patient will be seen in consultation of geriatry, otorhinolaryngology, pneumology, neuropsychology

SUMMARY:
Since December 2019, China and then the rest of the world have been affected by the rapid spread of a new coronavirus infection called SARS-CoV-2 (severe acute respiratory syndrome coronavirus), the clinical expression of which is called Covid-19 (Coronavirus Disease 2019).

It is estimated that around 20% of symptomatic patients will be severe enough to warrant hospitalization, of which around 5% will be in intensive care.

Organ damage is multiple in Covid infection: respiratory, digestive, renal, neurological, cardiovascular due to the infection or its care. There is also a psychological and social impact of the infection or of the care that should be measured.

In this context, investigator will assess the physical and psychological complaints of patients who have presented a severe form of SARS-CoV-2 infection.

The final objective being to identify the needs to offer follow-up adapted to this emerging pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for severe Covid-19 infection between March 1 and June 30, 2020 in a conventional unit, intensive care unit, at the Centre hospitalier du Mans and alive at the time of the investigation at 2 to 3 months
* Patient having given their express consent, after having received the research information letter upon discharge from hospital or having given their express consent after sending the information letter
* Age ≥ 18 years
* Patient having contracted a SARS-CoV-2 infection proved by RT-PCR and / or retrospective serology and / or a Covid-19 syndrome with suggestive chest scanner (during the period from March 1, 2020 to June 30, 2020)

Exclusion Criteria:

* Patient opposition to participate in the cohort
* Non-French speaking patient
* Patients who cannot read or write
* Patient subject to a protective measure
* Patient not affiliated to a social security or equivalent health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2022-06-11 (Estimated)

PRIMARY OUTCOMES:
Identify functionnal and psychosocial complaints | 3 months after last hospitalization
  the prevalence of functional complaints and psycho-social complaints (justifying additional investigations in patients hospitalized for Covid-19 infection 3 months maximum after discharge from hospital) will be assessed by questionnaire "Modified Medical Research Council"
Identify functionnal and psychosocial complaints | 3 months after last hospitalization
  the prevalence of functional complaints and psycho-social complaints (justifying additional investigations in patients hospitalized for Covid-19 infection 3 months maximum after discharge from hospital) will be assessed by questionnaire "Medical Outcome Study Short Form 36 (MOS SF-36)"
Identify functionnal and psychosocial complaints | 3 months after last hospitalization
  the prevalence of functional complaints and psycho-social complaints (justifying additional investigations in patients hospitalized for Covid-19 infection 3 months maximum after discharge from hospital) will be assessed by FRIED criteria
Identify functionnal and psychosocial complaints | 3 months after last hospitalization
  the prevalence of functional complaints and psycho-social complaints (justifying additional investigations in patients hospitalized for Covid-19 infection 3 months maximum after discharge from hospital) will be assessed by questionnaire "Hospital Anxiety and Depression Scale (HADS)"

SECONDARY OUTCOMES:
description of functionnal and psychosocial complaints | 3 months after last hospitalization
  complaints will be assessed by questionnaire "Modified Medical Research Council"
description of functionnal and psychosocial complaints | 3 months after last hospitalization
  complaints will be assessed by questionnaire "Medical Outcome Study Short Form 36 (MOS SF-36)"
description of functionnal and psychosocial complaints | 3 months after last hospitalization
  complaints will be assessed by FRIED criteria
description of functionnal and psychosocial complaints | 3 months after last hospitalization
  complaints will be assessed by questionnaire "Hospital Anxiety and Depression Scale (HADS)"
Identify the factors favoring the persistence of complaints | 3 months after last hospitalization
  Risk factors are defined according to age, concomitant treatment, comorbidities before hospitalization
Describe functional, neuropsychological and social complaints at a distance | 3 months after last hospitalization
  Complaints will be assessed by questionnaire"Modified Medical Research Council"
Describe functional, neuropsychological and social complaints at a distance | 3 months after last hospitalization
  Complaints will be assessed by questionnaire"Medical Outcome Study Short Form 36 (MOS SF-36)"
Describe functional, neuropsychological and social complaints at a distance | 3 months after last hospitalization
  Complaints will be assessed by FRIED criteria
Describe functional, neuropsychological and social complaints at a distance | 3 months after last hospitalization
  Complaints will be assessed by questionnaire "Hospital Anxiety and Depression Scale (HADS)"
Describe the needs for medical and surgical consultations after discharge from hospital | 3 months after last hospitalization
  Medical and surgical consultations after discharge will be measured as percentage
Describe the needs for neuropsychological support, dietetics, social assistance after discharge from hospital. | 3 months after last hospitalization
  neuropsychological support, dietetics, social assistance after discharge will be measured as percentage
Describe the factors of inequalities in access to care | 3 months after last hospitalization
  Describe the factors of inequalities in access to care and study their impact on the occurrence of a SARS-CoV-2 infection, its severity and the occurrence of a functional or psycho-social complaint.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier du Mans, Le Mans, France